CLINICAL TRIAL: NCT06667102
Title: Strategic and Interactive Signing Instruction (SISI): An Intervention Program to Support Sign Language Development in Deaf Children
Brief Title: Strategic and Interactive Signing Instruction
Acronym: SISI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UTennesseeKnoxville; R21DC021024 (NIH)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Teaching Behaviors; Sign Language Skills
Keywords: Sign language; Teacher training; Language deprivation
MeSH Terms: conditions — Sign Language

STUDY DESIGN:
Intervention Model Description: The PI will implement an experimental single case research design to track doses of SISI training and its efficacy in increasing teacher faithfulness to SISI.
  The PI will implement an experimental single case research design to identify causal relations between SISI and target sign language skills.
  The PI will implement a pre- and post- data to track deaf children's baseline growth in sign language skills prior to receiving SISI.
  The PI will implement a quasi-experimental study to identify the efficacy of SISI in improving deaf children's sign language skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Improving Teacher Fidelity to SISI (Experimental): A noncurrent multiple baseline design across teacher participants will be utilized to assess the extent of support required by teachers to become proficient in SISI implementation. In this study, the independent variable is the SISI training, and the dependent variable is teacher fidelity to the SISI program as measured by the SISI fidelity checklist.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Control and Experimental Groups: SISI Efficacy (Experimental): This pre- and post- study provides baseline data on deaf children's sign language development prior to receiving SISI. Additionally, each participating teacher will submit a recorded instructional unit showcasing their best methods for supporting sign language development. This provides a further layer of baseline analysis, allowing the PI to assess the instructional methods already in use prior to SISI professional development and implementation. Demographic data for both teachers and students will also be collected in preparation for the quasi-experiment study.
  Then, teachers will be assigned to either an experimental group, which will receive SISI professional development, or a control group that will continue with their usual teaching practices. In this quasi-experiment study, SISI's efficacy will be evaluated by comparing outcomes between the two groups.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Pre- and Post- Descriptive Study Data of Language Outcomes Children (Experimental): Up to 40 children from 4 classes will provide pre- and post-data in which they respond to a prompt in sign language on video.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Deaf Children's Language Growth (Experimental): Single case research design will provide robust day-to-day data of causal relations between SISI and sign language skills. Given teachers' high fidelity in SISI implementation, a noncurrent multiple baseline design across child participants will be applied to assess the extent of SISI improving deaf children's target sign language skills in a year. The independent variable of this study is the SISI implementation, which is used to improve the dependent variables which will be target sign language skills.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction

INTERVENTIONS:
Behavioral: Strategic and Interactive Signing Instruction — SISI centers on deaf children producing sign language compositions to communicate their messages with identified audiences, and teachers utilizing strategic and interactive approaches to bring attention to target sign language skills by consciously monitoring and manipulating language to create desired meanings grounded in socially shared understandings.

SUMMARY:
Strategic and interactive approaches driven by sociocultural, cognitive, and language theories have accumulated a large body of evidence documenting improvements in more complex oral and written language skills. Growing evidence demonstrates that more complex sign language skills positively predict literacy skills and may lead to improved health outcomes. This project involves new applications of theory-driven strategic and interactive approaches in an intervention program to target sign language development in deaf children between 5 and 8 years old who are at high risk of language delays.

DETAILED DESCRIPTION:
Deaf children who reach the age of eight without a foundation in language have longitudinal struggles in the areas of receptive and expressive language, working memory, executive functions, literacy and academic skills, and behavioral, mental, social, and physical health. The lack of intervention programs targeting sign language competencies during the critical period of development is a critical barrier to making progress in preventing or addressing language delays in deaf children. Strategic and interactive approaches driven by sociocultural, cognitive, and language theories have accumulated a large body of evidence documenting improvements in more complex oral and written language skills. Cross-linguistic transfers between oral and writing skills within and across first and second languages are well-established in the literature. Taking these factors into account in addition to growing evidence that sign language skills positively predict literacy skills and may lead to improved health outcomes, it is critical to systematically support deaf children's sign language competences as early as possible. To address the identified critical barrier to progress, these are the aims of this project: (1) develop Strategic and Interactive Signing Instruction (SISI), an intervention program to target the development of sign language skills in deaf children aged 5-8; (2) refine SISI training and implementation protocols; and (3) test the efficacy of SISI in improving deaf children's sign language skills. First, a SISI manual will be developed for standardization and consistency in training, implementation, and fidelity. The SISI manual will include: (a) descriptions of strategic and interactive approaches and their new applications to develop sign language skills, (b) SISI intervention protocols, (c) SISI fidelity checklist, and (d) list of sign language skills that are targeted in SISI. Second, an experimental study will be conducted to assess the extent of training and support required from teachers to become proficient in SISI implementation. Meanwhile, child progress in meeting their target sign language skills will be monitored formatively, and modifications may be made in an iterative design fashion to strengthen the intervention design. Third, another experimental study will be applied to assess the efficacy of SISI in improving deaf children's sign language skills. Findings will provide robust data on the mechanisms of successful training dose, intervention design and fidelity, and data collection protocols in preparation for subsequent R01 application involving a large randomized controlled trial with sufficient statistical power to further strengthen evidence of SISI in improving deaf children's sign language skills along with examinations of cross-linguistic interactions in the written form. This project is innovative in its new applications of theory-driven strategic and interactive approaches to target sign language development in deaf children.

ELIGIBILITY:
Inclusion Criteria:

* Deaf students in prekindergarten to 3rd grade classes
* Teachers of the deaf in prekindergarten to 3rd grade classes

Exclusion Criteria:

* Hearing students, deaf students aged 0-3 or 4th grade and beyond
* Non-teachers of the deaf or teachers of the deaf in 4th grade and beyond

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sign Language Skills | From enrollment to the end of treatment 9 academic months later.
  Deaf children's application of genre-based trait skills in sign language will be analyzed using rubrics adapted from the National Assessment of Educational Progress (NAEP) rubrics for standardized writing assessments.
Teaching Behaviors | From enrollment to the end of treatment 9 academic months later.
  Teachers' fidelity to SISI will be measured through the fidelity instrument.

SECONDARY OUTCOMES:
Written Language | From enrollment to the end of treatment 9 academic months later.
  Deaf children's application of genre-based trait skills in written language will be analyzed using the emergent writing stages and rubrics adapted from the National Assessment of Educational Progress (NAEP) rubrics for standardized writing assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The data from interventions in all four arms (two single case research designs and two baseline / quasi-experimental designs) will be shared in .csv files.
Supporting Information: CSR
Time Frame: IPD will be made available on 12/30/2026 with no end date.
Access Criteria: A researcher may access the IPD by contacting the principal investigator.